CLINICAL TRIAL: NCT04353791
Title: A Phase Ib/IIa, Randomized, Double Blind, Placebo Controlled, Multicenter Clinical Trial to Evaluate the Safety, Pharmacokinetics and Efficacy of Oral Treatment With OST-122 in Patients With Moderate to Severe Ulcerative Colitis
Brief Title: Study of OST-122 in Patients With Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oncostellae S.L (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-OST-122-02
Record Dates: First submitted 2020-03-24; First posted 2020-04-20 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-01

CONDITIONS: Ulcerative Colitis Chronic Moderate; Ulcerative Colitis Chronic Severe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm OST-122 (Active Comparator): 24 subjects will be randomized to receive OST-122 orally daily for 28 days
  Interventions: Drug: OST-122
- Control arm Placebo (Placebo Comparator): 8 subjects will be randomized to receive placebo orally daily for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OST-122 — Active dose
  Arms: Experimental arm OST-122
Drug: Placebo — Placebo
  Arms: Control arm Placebo

SUMMARY:
A Phase Ib/IIa to evaluate the safety and tolerability of oral treatment with OST-122 in patients with moderate to severe ulcerative colitis over 28 days. This trial will also explore pharmacokinetics (PK) profile and preliminary therapeutic efficacy associated with OST-122 through biomarker analysis and clinical, endoscopic and histologic assessments.

DETAILED DESCRIPTION:
OST-122 is an oral, gut-restricted and subtype-selective Jak3/Tyk2/Ark5 inhibitor for the local treatment of inflammatory bowel disease (IBD) including ulcerative colitis, Crohn's disease and, potentially, fibrotic lesions in Crohn's patients. The compound was well tolerated in a Phase 1 study in healthy volunteers and has been shown to be stable during the GI transit, while no significant plasma levels were detected. The gut-restricted PK profile of OST-122 lowers the risk of systemic toxicities inherent to other JAK inhibitors. In the current proof of concept study, the compound's safety, PK profile and trends of efficacy will be investigated in patients with moderate to severe ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent and capable of understanding and complying with the protocol;
2. Patients male and female ≥ 18 and ≤ 75 years at the time of consent;
3. Patient with previous diagnosis of ulcerative colitis: ulcerative proctitis, left-side ulcerative colitis or extensive/pancolitis (E1, E2 and E3 of Montreal Classification, respectively) established at least 3 months prior to screening and determined by standard clinical, endoscopic, and histological procedures;
4. Demonstrated inadequate response, loss of response, or intolerance to at least one of the following treatments including, aminosalicylates (ASAs), corticosteroids, immunosuppressants, anti-tumor necrosis factor (TNF)-α agents, integrin inhibitor or anti interleukin 12/23;
5. If the subject is currently receiving an oral aminosalicylate, he or she is eligible and can stay on that dose of aminosalicylate provided the dose has been stable for at least 1 week prior to screening;
6. If the subject is currently receiving an oral corticosteroid, he or she is eligible if the dose is equivalent to or less than prednisone 20 mg/day or beclomethasone dipropionate 5 mg/day and stable for at least 1 week prior to Screening visit;
7. Has an endoscopic Mayo subscore of ≥ 2 and a total Mayo score of 5-10 during screening;
8. Women who are not postmenopausal (at least 12 months) or surgically sterile must have a negative pregnancy test at screening and at the end of study and either abstain from sexual intercourse or use a highly effective method of birth control (double barrier) for the duration of the study and after 12 weeks after the last dose of study drug;
9. For men: agreement to remain abstinent or use contraceptive measures and agreement to refrain from donating sperm for the duration of the study and after 12 weeks from the last dose of study drug;
10. Availability for the entire study period, absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements; willingness to adhere to the protocol requirements, ability to cooperate adequately and to understand and follow the instructions of the physician or designee.

Exclusion Criteria:

1. Has fulminant colitis, toxic megacolon, primary sclerosing cholangitis, Crohn's disease, history of moderate to severe colitis-associated colonic dysplasia, active peptic ulcer disease;
2. Medications of exclusion:

   1. Topical mesalazine or steroids (i.e., enemas or suppositories) within the 7 days prior to Baseline visit
   2. Azathioprine, 6-mercaptopurine, or methotrexate within 10 days prior to Baseline visit
   3. Intravenous corticosteroids within the 14 days prior to Baseline visit
   4. Tofacitinib or any other JAK inhibitor within 14 days prior to Baseline visit
   5. Anti-diarrheal treatment within 14 days prior to Baseline visit
   6. Received cyclosporine, tacrolimus, mycophenolate mofetil, or thalidomide within 14 days prior to Baseline visit
   7. Adalimumab within the 14 days prior to Baseline visit
   8. Infliximab, golimumab, etanercept, vedolizumab, ustekinumab or certolizumab within the 14 days prior to Baseline visit
   9. NSAIDs on a daily basis from 7 days previous to Baseline visit. Low doses, without anti-inflammatory effect, to treat or prevent other diseases i.e.: ictus, cerebrovascular or cardiovascular diseases, among others; are permitted.
3. Has a current bacterial, parasitic, fungal, or viral infection;
4. Is positive for hepatitis A, B or C, HIV (Human Immunodeficiency Virus) or tuberculosis, as assessed by method available at each site;
5. Patient who has clinically significant diseases and/or infections captured in the medical history or evidence of clinically significant findings on physical examination and/or clinically significant ordinary laboratory evaluations (haematology, biochemistry, and urinalysis) or ECG;
6. Participated in another clinical trial of an investigational drug (or medical device) within 30 days prior to Baseline (or within 60 days prior to Baseline if investigational drug was a biologic product);
7. Demonstrated an inadequate response or loss of response to Tofacitinib or any other JAK inhibitor, with the exception of those patients who after a careful evaluation, the PI considers they may obtain a clinical benefit from the therapy;
8. Use of products, food supplements or medical devices, whose composition includes probiotics in the 1 month prior to Baseline visit;
9. Patient who has prior extensive colonic resection, subtotal or total colectomy or planned surgery for ulcerative colitis;
10. Patient who has past or present fistula or abdominal abscess;
11. Patient who is pregnant or lactating;
12. Inability to comply with study protocol, in opinion of the investigator;
13. History of alcohol, drug or chemical abuse within 6 months prior to Screening visit;
14. History of cancer within the last 5 years. Patients with local basal or squamous cell carcinoma of the skin that has been excised and is considered cured may be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of OST-122 administered for 28 days in subjects with active UC by assessing the number, severity, and type of adverse events | From baseline to end of the follow-up period
  Number and severity of AEs reported including Clinically Significant Changes in vital signs, physical examination, Laboratory Measurements, and ECGs.

SECONDARY OUTCOMES:
Cmax: Maximum plasma concentration for OST-122 | Day 1 and Day 28
  Pharmacokinetic analysis of OST-122 peak concentration in plasma (ng/ml) in every subject enrolled in this trial
Ctrough: Minimum plasma concentration for OST-122 | Day 1 and Day 28
  Pharmacokinetic analysis of OST-122 minimum concentration in plasma (ng/ml) in every subject enrolled in this trial
Tmax: Time to reach maximum plasma concentration (Cmax) for OST-122 | Day 1 and Day 28
  Pharmacokinetic analysis of OST-122 time (in hours) needed for OST-122 to reach the Cmax (peak concentration) in every subject enrolled in this trial
AUC: Area under the plasma-concentration time-curve | Day 1 and Day 28
  Pharmacokinetic analysis of OST-122 observed area under the plasma-concentration time-curve (ng · h / ml) in every subject enrolled in this trial
Percentage of subjects with improvement in Endoscopic Mayo Score | Day 0 and Day 28
  Study the effect of OST-122 or placebo in Endoscopic Mayo Score
  Subjects (%) with improvement of endoscopy subscore by ≥1 point Subjects (%) with endoscopy subscore of 0-1
Percentage of subjects with improvement in PRO-2 | Day 0, Day 7, Day 14, Day 21, Day 28
  Study the effect of OST-122 or placebo in PRO-2 [PRO-2: sum of the scores obtained in rectal bleeding and stool frequency (subscores 1+2 of the Mayo Score)]
  Subjects (%) with PRO-2 subscore of 0-1 Subjects (%) with improvement of PRO-2 subscore by ≥1 point Subjects (%) with improvement of rectal bleeding subscore by ≥1 point Subjects (%) with rectal bleeding subscore of 0-1 Subjects (%) with improvement of stool frequency subscore by ≥1 point Subjects (%) with stool frequency subscore of 0-1
Study the effect of OST-122 or placebo on faecal calprotectin levels | Day 1, Day 7, Day 14, Day 21, Day 28
  Change from baseline of faecal calprotectin (mg/kg) compared to placebo
Effect of OST-122 or placebo on serum C-reactive protein levels | Day 0, Day 14, Day 28
  Change from baseline of serum C-reactive protein (mg/L) compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Ascensión Heredia Rodríguez, PhD, Study Director — Oncostellae S.L
Locations (16):
- Spain (14):
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Reina Sofía, Córdoba
  - Hospital Universitari Doctor Josep Trueta, Girona
  - Hospital San Jorge, Huesca
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- Ukraine (2):
  - Medical and Diagnostic Center PE PMC "Acinus", Kropyvnytskyi
  - Medical Center "Ok!Clinic" of International Institute of Clinical Research LLC, Kyiv